CLINICAL TRIAL: NCT00999128
Title: An Open-Label, Two-Part Study to Determine the Relative Bioavailability of Capsule and Tablet Formulations of GDC-0941 and the Effect of Food and Proton Pump Inhibition on GDC-0941 Tablet Pharmacokinetics in Healthy Volunteers
Brief Title: A Study to Determine the Relative Bioavailability of Capsule and Tablet Formulations of GDC-0941 and the Effect of Food and Proton Pump Inhibition on GDC-0941 Tablet Pharmacokinetics in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GDC4740g
Record Dates: First submitted 2009-10-19; First posted 2009-10-21 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2010-02

CONDITIONS: Healthy Volunteers
Keywords: PI3K inhibitor; PI3 kinase; PI3 kinase inhibitor
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies | interventions — 2-(1H-indazol-4-yl)-6-(4-methanesulfonylpiperazin-1-ylmethyl)-4-morpholin-4-ylthieno(3,2-d)pyrimidine; Rabeprazole

ARMS (2):
- Part 1 (Experimental)
  Interventions: Drug: GDC-0941
- Part 2 (Experimental)
  Interventions: Drug: GDC-0941; Drug: rabeprazole

INTERVENTIONS:
Drug: GDC-0941 — Oral repeating dose
Drug: rabeprazole — Oral repeating dose
  Arms: Part 2

SUMMARY:
This is a Phase I, randomized, two-part, single-center pharmacokinetics (PK) study to assess the relative bioavailability of capsule and tablet formulations of GDC-0941 in the fasted state (Part 1) and to determine the effect of food and proton pump inhibition on the PK of the tablet formulation of GDC-0941 (Part 2). Approximately 18 subjects will be enrolled in Part 1 and up to 32 subjects will be enrolled in Part 2. Subjects who participate in Part 1 are not eligible to participate in Part 2.

ELIGIBILITY:
Inclusion Criteria

* Male or female, between 18 and 65 years of age, inclusive (Part 1 only)
* Male or female, between 18 and 45 years of age, inclusive (Part 2 only)
* In good health, as determined by no clinically significant findings from medical history, 12-lead electrocardiogram (ECG), and vital signs assessment
* Body Mass Index (BMI) between 18-30 kg/m^2 inclusive, with a body weight >50 kg
* Clinical laboratory evaluations within the reference range for the test laboratory
* Negative test for selected drugs of abuse at screening (does not include alcohol) and at check-in (does include alcohol)
* Negative HIV, hepatitis B surface antigen (HBsAg), and hepatitis C virus antibody screens
* Agreement to use an effective form of contraception for the duration of the study

Exclusion Criteria

* History or clinical manifestations of significant metabolic (including type 1 and 2 diabetes), hepatic, renal, hematological, pulmonary, cardiovascular, endocrine, gastrointestinal, urological, neurological, psychiatric disorders, or cancer
* History of inflammatory arthritis
* History of symptomatic hypotension
* History of severe physical injury, direct impact trauma, or neurological trauma within a specified timeframe prior to Day 1
* History of seizure disorders
* History of bipolar or major depressive disorder
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (exceptions: appendectomy, hernia repair, and/or cholecystectomy)
* History or presence of an abnormal ECG
* Subjects with a history of ventricular dysrhythmias or with risk factors for ventricular dysrhythmias
* History of alcoholism, drug abuse, or drug addiction
* Use of any nicotine-containing or nicotine-replacement products within a specified timeframe prior to Day 1
* Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within a specified timeframe prior to Day 1
* Use of any prescription medications/products within a specified timeframe prior to Day 1 (exceptions: hormone replacement therapy [HRT], oral, implantable, or transdermal contraception)
* Receipt of any vaccination or immunization within a specified timeframe prior to Day 1
* Use of proton pump inhibitors or H2-receptor antagonists within a specified timeframe prior to Day 1
* Known hypersensitivity to rabeprazole or any of its components, or to derived products of benzimidazoles
* Use of any over-the-counter (OTC), non-prescription preparations within a specified timeframe prior to Day 1
* Use of alcohol-containing, grapefruit-containing, or caffeine-containing foods or beverages within a specified timeframe prior to Day 1
* Poor peripheral venous access
* Donation of blood or plasma within a specified timeframe prior to Day 1
* Receipt of blood products within a specified timeframe prior to Day 1
* Vegetarians who are unable to consume a high-fat meal
* Women who are pregnant or nursing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-10-26 (Actual); Primary Completion 2010-02-26 (Actual); Study Completion 2010-02-26 (Actual)

PRIMARY OUTCOMES:
Incidence, nature, and severity of adverse events | Through study completion or early study discontinuation
PK parameters of GDC-0941 (total exposure, maximum and minimum plasma concentration) | Following administration of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Scott Holden, M.D., Study Director — Genentech, Inc.
Locations (1):
- Genentech Trial Information Support, South San Francisco, California, United States